CLINICAL TRIAL: NCT05147194
Title: The Effects of Trimetazidine on Diabetic Nephropathy
Brief Title: The Effects of TMZ on Diabetic Nephropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-DN-TMZ
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Trimetazidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Blank group
- Trimetazidine group (Experimental): The participates received treatments of trimetazidine
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — Oral，35mg bid
  Arms: Trimetazidine group

SUMMARY:
With the improvement of people's living standard, the prevalence of Diabetes is increasing year by year. In present, 350 million people worldwide are suffering from diabetes, and by 2035, there will be as high as 600 million. Diabetes causes a variety of complications, including diabetic nephropathy, which is one of the most common complications of Diabetes. Diabetic nephropathy is a microvascular complication of diabetes. Microalbuminuria and glomerular filtration rate decrease are the main manifestation. Even more, it can progress to end-stage renal changes. Data showed that diabetic nephropathy accounts for about 40% of patients with end-stage renal disease receiving renal replacement therapy.

However, the treatment of diabetic nephropathy is still lacking. In the past 40 years, few drugs have been proven to ameliorate the progression of diabetic nephropathy. Even though, the renal function of a large number of diabetic nephropathy patients is gradually deteriorating. Therefore, it is urgent to find a therapeutic drug that acts on different targets.

Trimetazidine is a piperazine derivative. It is mainly used in the treatment of stable angina pectoris. Its safety has been well verified. In recent years, the role of trimetazidine in acute renal damage has been widely reported. A large number of studies have shown that trimetazidine can reduce the effect of contrast agent on renal function and reduce the incidence of contrast nephropathy. There fore, Trimetazidine is a promising drug for delaying the progression of diabetic nephropathy.

DETAILED DESCRIPTION:
In the present study, there will be 2 groups last for 6 months. One is the control group, who will not receive trimetazidine and the another is the trimetazidine group, who will receive the treatment of trimetazidine, 35mg bid orally.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age;
2. Type 2 diabetes mellitus;
3. EGFR ≥30 to <90 ml/min/1.73 m2;
4. Urinary albumin creatinine ratio (UACR) ≥ 30 mg/g;

Exclusion Criteria:

1. Women who are already pregnant or planning to become pregnant;
2. SBP >180mmHg and/or DBP >110mmHg;
3. UACR ≥ 3000 mg/g
4. Other non-diabetic renal diseases (such as polycystic kidney disease, lupus nephritis, ANCA-associated vasculitis, etc.);
5. NYHA cardiac function grade III or above
6. Those who have a history of cancer or are currently suffering from cancer;
7. Receiving immunosuppressant, cytotoxic or other immunosuppressive therapy in the first 6 months;
8. Patients with acute coronary syndrome, acute cardiac insufficiency or severe cerebrovascular disease in the previous month;
9. Patients refused to comply with the requirements of the study to complete the study;
10. In the investigator's judgment, the patient is unable to complete the study or comply with the requirements of the study (for management reasons or other reasons);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of UACR levels at 6 months to baseline UACR | 6 month
  UACR(6 M)/UACR（base）

SECONDARY OUTCOMES:
Serum creatinine | 6 month
  Serum creatinine
24h urine protein level | 6 month
  24h urine protein level
Proportion of patients with UACR>300 mg/g in the population at 6 months | 6 month
  Proportion of patients with UACR>300 mg/g in the population at 6 months
Proportion of patients with UACR >30mg/g and <300 mg/g in the population at 6 months | 6 month
  Proportion of patients with UACR >30mg/g and <300 mg/g in the population at 6 months
Ratio of UACR levels at 3 months to baseline UACR | 3 month
  Ratio of UACR levels at 3 months to baseline UACR
Ratio of UACR levels at 1 months to baseline UACR | 1 month
  Ratio of UACR levels at 1 months to baseline UACR